CLINICAL TRIAL: NCT01188096
Title: A Phase II Trial of Poly-ICLC in the Management of Recurrent Pediatric Low Grade Gliomas
Brief Title: A Trial of Poly-ICLC in the Management of Recurrent Pediatric Low Grade Gliomas
Acronym: Poly-ICLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Poly ICLC; 004385 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Results first posted 2023-04-03 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Brain Tumors
Keywords: glioma; pediatrics; cancer; brain tumor; low grade glioma
MeSH Terms: conditions — Brain Neoplasms; Glioma; Neoplasms | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Poly ICLC (Experimental): Children will receive poly-ICLC 20 mcg/kg twice weekly intramuscular injection (IM). The first 2 doses will be administered in the clinic under supervision.
  Interventions: Drug: Poly ICLC

INTERVENTIONS:
Drug: Poly ICLC — Children will receive poly-ICLC 20 mcg/kg twice weekly IM (using Monday/Wednesday schedule if possible). The first 2 doses will be administered in the clinic under supervision.

SUMMARY:
This study is for patients up to 21 years of age who have a tumor called a low grade glioma of the central nervous system (brain and spinal cord). The tumor has grown despite attempts to control it with chemotherapy or radiation. Low grade gliomas are a group of tumors that tend to grow slowly and could be cured if every bit of the tumor were surgically removed. These tumors are called Grade I or II astrocytomas.

These tumors often grow in parts of the brain that prevent total removal without devastating neurologic complications or death. Although some low grade gliomas never grow, most will and are treated with either chemotherapy or radiation. There is good data showing that the growth of most low grade gliomas can be controlled with chemotherapy or radiation. However, some low grade gliomas in children and young adults grow despite these treatments. Poly-ICLC is a new drug that has been used safely in children and adults with different types of brain tumors. Earlier studies showed that this drug worked better for children and young adults with low grade gliomas than for children with more aggressive brain tumors. The main purpose of this study is to use Poly-ICLC treatment in a larger number of patients to see how well it works and how many side effects occur.

As Poly-ICLC is not FDA approved, this study is authorized to use it under Investigational New Drug (IND)# 43984, held by Oncovir.

Subjects will get injections of Poly-ICLC into muscle two times weekly. The first treatments will be given in the clinic so allergic or other severe reactions, if any, can be monitored. If subjects tolerate the injections and don't have a severe reaction, then the rest of the injections will be given at home. Subjects/caregivers will be trained to give injections.

Treatment will last for about 2 years. Subjects may stay on treatment for longer than 2 years if their tumor shrinks in response to the injections, if study doctors think it is safe, if subjects want to remain on treatment, and if Poly-ICLC is available.

Risks: Poly-ICLC has been used safely in children and adults at the dose used in this study, and at higher doses. Frequently seen side effects include irritation of the skin at the injection site and mild flu-like symptoms. These are usually relieved or avoided by use of over-the-counter medicines like acetaminophen (Tylenol).

DETAILED DESCRIPTION:
Background/Rationale The incidence of primary pediatric brain tumors in the United States is about 1500 per year. Brain tumors are the most common solid tumor diagnosed in childhood and thus account for significant childhood mortality in the United States. Low-grade astrocytomas and gliomas are the most common type of brain tumor of childhood (36% of childhood brain tumors). These tumors encompass a heterogeneous assortment of histological subtypes including: fibrillary, protoplasmic, gemistocytic, and mixed variants. Pilocytic astrocytomas, pleomorphic xanthoastrocytomas and subependymal giant cell astrocytomas are also included. Furthermore, in young children there are some unique rare entities that behave like low-grade tumors, including infantile desmoplastic gangliogliomas, and desmoplastic astrocytomas. Although children with low-grade astrocytomas often survive many years after conventional treatment with surgery and sometimes radiotherapy, some children will not fare as well. These tumors constitute a heterogeneous group because of differing locations within the brain and varying biological behavior of different subtypes. For those where total excision is possible, such as cerebellar astrocytomas, prognosis is excellent with over 90% ten-year survival rates with surgical excision alone. In contrast, survival rates in children with cerebral or diencephalic tumors are 40-70% at five years with irradiation, but decline to 11-50% at 10 years. Some tumors however may be unresectable/partially resectable, and radiation can have undesirable side effects in young children. While the most significant intellectual deficits occur in young children less than 5 years treated with cranial irradiation, the deficits recognized even in young adults warrant extending the age to 10 years for avoiding radiation. Chemotherapy regimens are used for high-risk patients (progressive tumor, residual tumor) as a means to avoid or delay radiation in young patients, but side effects of chemotherapy are frequently reported.

Newer forms of effective treatment that will have lesser side effects are much needed in childhood brain tumors especially low-grade gliomas. We propose to study the efficacy and toxicity of poly-ICLC, a biological response modifier in children with low-grade gliomas.

PROTEOMICS

Current diagnostic and therapeutic monitoring of brain tumor patients are significantly hindered due to limited understanding of brain tumor biology and response to therapy. The majority of central nervous system (CNS) tumors cannot be identified or followed by expression of serum or Cerebrospinal fluid (CSF) markers. However, if available, such markers would be highly desirable and could be used to:

* Detect minimal residual disease
* Predict response to specific targeted therapies
* Predict or anticipate tumor progression
* Distinguish tumor recurrence from post surgical changes or post-radiation changes on neuro-imaging
* Augment current histopathologic classification systems
* Improve current clinical and pathological treatment stratification schemata
* Assess efficacy of and tumor response to specific biologic targeted therapies that may not impact tumor size as a primary tumor endpoint (e.g., small molecule inhibitors or anti-angiogenic strategies) While such markers would be useful to prognosticate, monitor and treat all CNS tumors, its use in glial tumors including recurrent low grade astrocytomas is critical since these tumors are often biopsied at presentation, but not at recurrence. Often these tumors are not amenable complete resection or biopsy due to the eloquence of brain tissue they infiltrate (e.g., optic pathway, brainstem or hypothalamic gliomas), or the blood vessels that they encase.

CNS biologic material in CSF Glial tumors tend to disseminate locally along white matter tracts rather than through sub-arachnoid seeding. Dissemination of low grade gliomas along the sub-arachnoid space has been reported in children with low grade gliomas. Even focal tumors are frequently adjacent to CSF pathways (e.g., intrapeduncular fossa, third and fourth ventricles) resulting in direct contact between tumor tissue and spinal fluid. Yet examination of CSF cytology for these tumors is not standard. Given limitations of identifying tumor cells in the CSF, methodologies that could improve our understanding of CNS tumors of all types are needed. This would provide a significant improvement in currently available knowledge about the biology of these tumors, and could elucidate potential therapeutic avenues.

Proteomics, a relatively new area of research whereby total protein complement of a tissue compartment is analyzed, has successfully been used to identify novel biomarkers in solid tumors. Because proteins are effectors of all cellular functions, their measurement should represent the most direct means of cellular characterization and hence tumor biology. Because cells and their environment exist in an integrated state, it has been possible to interrogate the proteins of extra-cellular compartments to assess the presence and impact of tumor cells. This has been done primarily using serum or plasma to establish a method of screening for the presence of low stage tumors. An analogous extra-cellular compartment for use in brain tumors would be cerebrospinal fluid (CSF). It circulates throughout the CNS and exchanges proteins with the extra-cellular fluid of the brain and spinal cord.

CSF is continuously created and reabsorbed, providing a real time steady state proteome. Unlike serum, which contains a highly complex protein mixture ranging from very low abundance proteins in the 10-30 pg/mL range to very abundant proteins in the 35-55 mg/mL range, CSF contains a less complex protein mixture.

Therefore, the CSF is more likely to contain higher relative concentrations of tumor-specific proteins (higher signal to noise ratio) than serum. Taken together this makes CSF and attractive alternative to serum for detection of brain tumor related biomarkers. Unlike leukemia and many solid tumors outside the CNS, where serial biopsies are readily performed, tumors of the CNS are not easily accessible other than at the time of initial or repeat resection or biopsy. While studies on these samples provide important findings regarding tumor biology, serial analyses during treatment are not reasonable. By contrast, the CSF of tumor patients can be more readily sampled in most pediatric patients. With the development of proteomic technology, investigation of tumor related signals at the time of diagnosis through treatment, and then in remission and/or at the time of recurrence or progression is possible.

While CSF for seeding tumors is readily available and routinely obtained for cytology, the systematic evaluation of the proteins within these samples could be of considerable scientific importance. In addition to identifying potential makers of disease or response to therapy, the glycosylation and phosphorylation status of many proteins can also be evaluated. Studies in tumor tissue show that such information reveals activity of different enzymes that correlate with treatment response or progression of leptomeningeal metastases.

Proteomics CSF proteomics has been applied to many neurological disorders including Alzheimer's disease, amyotrophic lateral sclerosis, multiple sclerosis, acute brain injury and Creutzfeldt-Jakob disease.

Reports of its use in neuro-oncology are limited, but demonstrate the potential of this technology to effectively identify tumor biomarkers. One study used two dimensional polyacrylamide (2-D) gel electrophoresis to measure the relative quantities of two pre-selected markers, proto-oncogene protein (N-Myc) and Intracranial atherosclerotic disease (l-CaD), in the CSF of brain tumor patients. CSF proteomics using 2-D gel electrophoresis in combination with mass spectroscopy and cleavable isotope Coded Affinity Tag (cICAT) was used to evaluate 60 samples of CSF and tumor cyst fluid taken from adults with brain tumors and non-neoplastic controls. These techniques were used to find a panel of proteins differentially expressed in lower vs. higher-grade gliomas. Findings were confirmed using Western Blot analysis probing for eight selected proteins based on implied role in gliomagenesis and availability of antibodies. This report, which has been accepted for publication pending revisions, identified 21 potential CSF biomarkers for astrocytoma.

As mentioned above, there is evidence that gliomas disseminate through the subarachnoid space. Currently there are several consortia actively studying protein expression in the spinal fluid of children with malignant glial and embryonal tumors. Proteins interrogated in these protocols include those involved with angiogenesis and neovascularity, those involved in tumor growth and migration (Secreted protein with acidic and cysteine rich domains (SPARC), attractin). There is no consortium actively collecting spinal fluid sample in children with lower grade tumors. A secondary goal of this study is to examine these proteins in the CSF of children with low grade gliomas who have tumor progression. Comparison of CSF protein expression of in high grade and low grade tumors is likely to help identify biological markers specific for tumor progression, or for tumor pathology.

ELIGIBILITY:
Inclusion Criteria:

* Age:Patients must be between 0 - 21 years of age when registered on this protocol.
* Diagnosis:Patients must have pathologically confirmed low grade glioma with histologic subtypes interpreted as World Health Organization (WHO) grade I and II including:
* juvenile pilocytic astrocytoma (JPA)
* pleomorphic JPA
* diffuse astrocytoma (fibrillary, gemistocytic, giant cell, or pleomorphic xanthoastrocytoma)
* low grade oligoastrocytoma
* low grade oligodendroglioma
* low grade glioma not otherwise specified (NOS) Tumors of all regions of the CNS, with appropriate histology are eligible for study. However patients with tumors intrinsic to the optic nerve and involvement of the optic nerve cannot be biopsied/resected are eligible without histological confirmation.

Patients with neurofibromatosis type 1(NF1) are also eligible.

Patients must have demonstrated either tumor progression or recurrence by radiographic criteria and/or clinical criteria as defined below:

1. Patients with progressive non-resectable disease regardless of location in the brain or spine are eligible for this study. Patients with evidence of leptomeningeal dissemination are eligible for this study. Patients do not require biopsy/histologic confirmation at the time of progression or relapse.
2. Radiographic progression is defined as >40% increase in the product of the three perpendicular diameters of initial tumor relative to the initial baseline measurement - length (L)x width (W) x transverse (T) (current scan) > 1.4 x L x W x T (initial scan), or the development of any new sites of disease independent of the response of the initial tumor. See section 7.1.2 for methodology for tumor measurement.
3. Post radiation changes are often seen on post-treatment imaging studies, so that classification of a patient as having progressive disease may require several serial MRI's if the child has received radiation within the preceding 12 months.
4. Tumor volume includes the entire tumor volume seen on gadolinium enhanced T1 MRI plus non-enhancing abnormality seen on T2 or FLAIR.
5. All tumor cysts will be included in the tumor volume
6. Clinical progression without radiographic progression includes children with optic pathway gliomas who demonstrate sustained decrease in visual fields and/or acuity in three serial vision examinations. Each of the vision examinations must be performed >2 weeks apart.
7. Children with previously negative cerebrospinal fluid (CSF) cytology who show evidence of tumor cells in fluid obtained by lumbar puncture can be designated as having progressive disease in the absence of radiographic evidence of progression.

Measurable disease: Patients must have measurable disease documented by radiographic criteria prior to enrollment.

Performance Level and Life Expectancy:Patients must have a performance status of > 50% (Appendix I). Use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age. Patients must have a life expectancy of ≥ 8 weeks.

Prior Therapy:Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study and meet time restrictions from end of prior therapy as stated below:

1. Myelosuppressive chemotherapy patients must have received the last dose of myelosuppressive therapy at least 3 weeks prior to study registration or at least 6 weeks if nitrosourea.
2. Investigational / Biological agent: Patient must have received the last dose of other investigational or biological agent >7 days prior to study registration
3. Radiation therapy (XRT): Patients must be ≥ 8 weeks since the completion of radiation therapy.
4. Study specific limitations on prior therapy: There is no limit on the number of prior treatment regimens or received doses of radiation therapy.
5. Growth factor(s): Must not have received any hematopoetic growth factors within 7 days of study entry or 21 days for neulasta.
6. Prior Surgery: Must be ≥ 2 weeks from prior surgery.
7. Steroids: Must be on a stable steroid dose for 7 days prior to study entry.

Organ Function Requirements:All patients must have adequate organ function defined as:

Hematologic Function:

1. Hemoglobin: > 8.0 gm/dl
2. Absolute neutrophil count (ANC): > 750/mm3 Must be at least 7days after last dose of growth factor
3. Platelet Count: > 50,000 (transfusion independent; ≥ 7 days from last transfusion)

Renal Function:

Serum creatinine ≤ 2 x normal for age (see below) or Creatinine clearance/Glomerular filtration rate (GFR) > 60 cc/min/1.73 m2 [Urine Creatinine (mg/dL)][Volume collected (ml)]/[Serum Creatinine 9mg/dL)][Hours x 60]

Age (years) Maximum Serum Creatinine (mg/dL)

≤ 5 0.8 > 5 & ≤ 10 1.0 > 10 & ≤ 15 1.2 > 15 1.5

Liver Function:

1. Total bilirubin < 1.5 x Upper limit of Normal (ULN) for age, AND
2. alanine transaminase (ALT) < 2.5x ULN
3. aspartate aminotransferase (AST) < 2.5x ULN

Pulmonary Function:

No evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry ≥ 94% if there is clinical indication for determination.

Coagulation Function:

Normal prothrombin time (PT) and Partial thromboplastin time (PTT) at enrollment per institutional range

Reproductive Function:Due to potential teratogenic effects of (poly-ICLC), negative serum beta-human chorionic gonadotropin (HCG) in females, and use of effective contraception in males and females of childbearing potential, IS REQUIRED.

Exclusion Criteria:

* Pregnant or lactating females. Women of childbearing age will agree to use contraception during the protocol.
* Patients receiving other experimental immunotherapy.
* Patients may not have fever (38.50C) within 7 days of enrollment.
* No concurrent XRT or chemotherapy is allowed.
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2010-08; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Durden, MD, Ph.D., Principal Investigator — University of California Medical Center
Locations (2):
- United States (2):
  - RADY Children's Hospital, San Diego, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neuro-Oncology, Volume 20, Issue suppl_6, November 2018, Page vi201, https://doi.org/10.1093/neuonc/noy148.833 Published: 05 November 2018
- See also: clinical trials database — http://www.choa.org/default.aspx?id=1957
- See also: Children's Healthcare of Atlanta — http://www.choa.org/
- See also: Emory University — http://www.emory.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Poly ICLC
Started | 23
Completed | 17
Not Completed | 6
Not completed — progression of disease | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Poly ICLC
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.17 (4.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Percentage with no progression of disease by MRI 3D Macdonald criteria. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 6 months
Measure: Number; unit: percentage of no progression
Arm/Group | Poly ICLC
Number analyzed (Participants) | 23
percentage of no progression | 70

2. Secondary Outcome: Overall Response Rate
Description: Tumor assessments are to be performed per Modified McDonald's criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar criteria for the Modified Mcdonald's Criteria, as accurate and appropriate.
Time Frame: at 6 months following start treatment with study drug
Measure: Number; unit: percentage of response
Arm/Group | Poly ICLC
Number analyzed (Participants) | 23
percentage of response | 74

3. Secondary Outcome: Overall Response Rate
Description: Tumor assessments are to be performed per 3D measurements. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar criteria for the Modified Mcdonald's Criteria, as accurate and appropriate.
Time Frame: at 2 years after start of treatment with study drug
Measure: Number; unit: percentage of response
Arm/Group | Poly ICLC
Number analyzed (Participants) | 23
percentage of response | 8.6

4. Secondary Outcome: Overall Survival Rate
Time Frame: month 6, 24 months
Measure: Number; unit: percentage of survival
Arm/Group | Poly ICLC
Number analyzed (Participants) | 23
percentage of survival
  Month 6 | 100
  Year 2 | 100

5. Other Pre Specified Outcome: Toxicity Associated With Treatment With Poly-ICLC
Description: in pediatric patients with recurrent low grade gliomas
Time Frame: month 6, 24 months
Population: collected during the study as AEs/SAEs and is reflected this way in the record
Arm/Group | Poly ICLC
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: The Effect of Treatment With Poly-ICLC on the Signaling Pathways Controlling Apoptosis in Low Grade Glioma Tumor Cells.
Time Frame: month 6, 24 months
Population: Outcome data was not collected and in the course of the study the outcome was not considered primary or secondary.
Arm/Group | Poly ICLC
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Surrogate Markers of Tumor Response and Progression Can be Identified in the Serum
Description: See if markers can be identified in the serum of patients with recurrent low grade gliomas treated with poly-ICLC.
Time Frame: month 6, 24 months
Population: Outcome data was not collected; and in the course of the study the outcome was not considered primary or secondary
Arm/Group | Poly ICLC
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Surrogate Markers of Tumor Response and Progression Peripheral Blood Mononuclear Cells (PBMC)
Description: Look for presence of markers in PBMC and/or cerebrospinal fluid of patients with recurrent low grade gliomas treated with poly-ICLC.
Time Frame: month 6, 24 months
Population: Outcome data was not collected; and in the course of the study the outcome was not considered primary or secondary
Arm/Group | Poly ICLC
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Surrogate Markers of Tumor Response and Progression--Cerebrospinal Fluid
Description: Look for presence of markers in cerebrospinal fluid of patients with recurrent low grade gliomas treated with poly-ICLC.
Time Frame: month 6, 24 months
Population: Outcome data was not collected; and in the course of the study the outcome was not considered primary or secondary
Arm/Group | Poly ICLC
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: from baseline through year 2
Arm/Group | Poly ICLC
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 5/23
Other Adverse Events (participants affected / at risk) | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poly ICLC (N=23)
Dehydration (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (1)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (1)
Stroke Intracranial Hemorrhage (Cardiac disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1)
Kidney Stone (Renal and urinary disorders) | 1 (1)
Adjustment of anti-seizure medications (General disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poly ICLC (N=23)
Anorexia (Gastrointestinal disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Bronchial Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
aspartate transferase (AST) Increase (Blood and lymphatic system disorders) | 6 (10)
Alanine transaminase (ALT) Increase (Blood and lymphatic system disorders) | 10 (23)
blood urea nitrogen (BUN) Increase (Blood and lymphatic system disorders) | 1 (1)
Bilirubin Increase (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (10)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (rash) (Skin and subcutaneous tissue disorders) | 1 (1)
Alkaline Phosphatase Increase (Blood and lymphatic system disorders) | 3 (3)
activated partial thromboplastin time (aPTT) Prolonged (Blood and lymphatic system disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (6)
Decreased absolute neutrophil count (ANC) (Blood and lymphatic system disorders) | 13 (35)
Creatinine Increase (Blood and lymphatic system disorders) | 2 (2)
Decreased Phosphate (Blood and lymphatic system disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2)
Decreased Platelet (Blood and lymphatic system disorders) | 3 (4)
Chills (General disorders) | 1 (1)
Decreased Visual Acuity Left Eye (Eye disorders) | 1 (1)
Decreased Visual Acuity Right Eye (Eye disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Genetic Disorder Neurofibromatosis type I (NFI) (Nervous system disorders) | 1 (1)
Faint (General disorders) | 1 (1)
Ear Infection (Ear and labyrinth disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
White Blood Cell (WBC) Decrease (Blood and lymphatic system disorders) | 12 (33)
Elevated aspartate aminotransferase (AST) (Blood and lymphatic system disorders) | 3 (5)
Elevated blood urea nitrogen (BUN) (Blood and lymphatic system disorders) | 1 (1)
Dry Eye (Eye disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Lymphocyte Decrease (Blood and lymphatic system disorders) | 15 (27)
Fever (General disorders) | 11 (20)
Headache (Nervous system disorders) | 6 (6)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 11 (28)
Hand Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypernatremia (Blood and lymphatic system disorders) | 3 (3)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hypoglycemia (Blood and lymphatic system disorders) | 3 (3)
Hypocalcemia (Blood and lymphatic system disorders) | 7 (21)
Hyperglycemia (Blood and lymphatic system disorders) | 2 (5)
Hypophosphatemia (Blood and lymphatic system disorders) | 11 (23)
Hyponatremia (Blood and lymphatic system disorders) | 3 (6)
Hypokalemia (Blood and lymphatic system disorders) | 2 (3)
Insomnia (General disorders) | 1 (2)
Motor Neuropathy (Nervous system disorders) | 1 (1)
Nystagmus (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Muscle soreness at Injection Site (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Middle Ear Inflammation (Ear and labyrinth disorders) | 1 (1)
Injection Site Pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Kidney Infection (Renal and urinary disorders) | 1 (1)
Pink Eye (Eye disorders) | 1 (1)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Lymphocyte (Blood and lymphatic system disorders) | 2 (3)
Optic Nerve Disorder (Left Esotropia) (Eye disorders) | 1 (1)
Optic Nerve Pallor (Eye disorders) | 1 (1)
low back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Obesity (General disorders) | 1 (1)
left knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spasticity (Musculoskeletal and connective tissue disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Weight Loss (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore arm (Musculoskeletal and connective tissue disorders) | 1 (3)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Platelet Count Increased (Blood and lymphatic system disorders) | 1 (1)
Renal Calculi (Renal and urinary disorders) | 1 (1)
Vaginal Infection (Reproductive system and breast disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-05-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT01188096/Prot_SAP_000.pdf
  • Informed Consent Form (2012-10-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT01188096/ICF_001.pdf